CLINICAL TRIAL: NCT02932462
Title: A Randomized, Double-Blind, Vehicle-Controlled, Parallel-Design, Multiple-Site, Phase III Clinical Study to Evaluate the Efficacy and Safety of DSXS 1535 in Patients With Mild to Severe Scalp Psoriasis
Brief Title: Study to Evaluate Efficacy and Safety of the Topical Product in Patients With Mild to Severe Scalp Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DSXS 1535
Record Dates: First submitted 2016-10-08; First posted 2016-10-13 (Estimated); Results first posted 2018-12-06 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-11

CONDITIONS: Scalp Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DSXS 1535 (Experimental): DSXS 1535 topical product
  Interventions: Drug: DSXS
- Placebo (Placebo Comparator): Vehicle
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DSXS — topical product
  Other Names: DSXS 1535
  Arms: DSXS 1535
Drug: Placebo — topical product
  Other Names: vehicle
  Arms: Placebo

SUMMARY:
A Randomized Double-Blind, Vehicle-Controlled, Parallel Design, Multiple-Site, Phase III Clinical Study

DETAILED DESCRIPTION:
This randomized, double-blind, vehicle-controlled, parallel-group multiple-site study is designed to evaluate the therapeutic efficacy and safety of the investigational product, DSXS 1535 product, for the treatment of mild to severe scalp psoriasis

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of mild to severe plaque psoriasis of the scalp, defined by an Investigator's Global Assessment (IGA) score of at least 2 at baseline/randomization

Exclusion Criteria:

* Patients whose scalp psoriasis necessitates systemic or other concomitant topical therapies during the study (concomitant treatment of body psoriasis with over the counter topical products including emollients, is allowed).
* Patient has a scalp skin condition that would interfere with the diagnosis or assessment of plaque psoriasis of the scalp (e.g., seborrheic dermatitis, eczema, cutaneous T-cell lymphoma, or other forms of psoriasis including guttate, inverse, pustular or erythrodermic psoriasis)
* Presence of pigmentation, extensive scarring, pigmented lesions, or sunburn in the treatment areas that could interfere with the rating of efficacy parameters, including planned extensive exposure to sunlight during the study.
* History of psoriasis unresponsive to topical treatments.
* Current immunosuppression or history of organ transplant.
* Patients who have a history of or current diagnosis of glaucoma.
* Patients who have had surgery on the eyes or eyelids within 1 month before baseline or plan to have eye or eyelid surgery during the study.
* Patients with active infection (including but not limited to bacterial, fungal and viral infection) and/or open wounds on the entire head and neck area.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 373 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2017-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novum Pharmaceutical Research Services, Study Chair — http://www.novumprs.com/contact; Natalie Yantovskiy, Study Director — Taro Pharmaceuticals USA Inc.

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DSXS 1535 | Placebo
Started | 184 | 189
Completed | 177 | 176
Not Completed | 7 | 13
Not completed — Adverse Event | 1 | 2
Not completed — Lost to Follow-up | 4 | 1
Not completed — Protocol Violation | 0 | 5
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Non-Compliance With Study Drug | 0 | 1
Not completed — Progressive Disease | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DSXS 1535 | Placebo | Total
Number analyzed (Participants) | 183 | 189 | 372
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (17.2) | 48.1 (17.3) | 48.1 (17.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 118 | 225
  Male | 76 | 71 | 147
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 77 | 85 | 162
  Not Hispanic or Latino | 106 | 104 | 210
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 5 | 4 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 17 | 14 | 31
  White | 159 | 165 | 324
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 4 | 5
Percent Scalp Affected [Mean (Standard Deviation); unit: percent] | 32.4 (26.6) | 33.5 (25.3) | 33.0 (25.9)
Number of months and/or years patient has suffered from symptoms caused by scalp psoriasis [Count of Participants; unit: Participants]
  <= 3 Months | 2 | 2 | 4
  >3 Months And <= 6 Months | 1 | 1 | 2
  > 6 Months And <= 1 Year | 8 | 11 | 19
  > 1 Year And <= 3 Years | 27 | 29 | 56
  > 3 Years And <= 5 Years | 29 | 28 | 57
  > 5 Years | 116 | 118 | 234

OUTCOME MEASURES:

1. Primary Outcome: Clinical Success in Patients With Moderate and Severe Scalp Psoriasis
Description: IGA score of 0 (clear) or 1 (almost clear) with at least a 2 grades reduction from baseline
Time Frame: from baseline to study day 29
Population: Patients with moderate and severe scalp psoriasis (primary analysis 1)
Measure: Count of Participants; unit: Participants
Arm/Group | DSXS 1535 | Placebo
Number analyzed (Participants) | 106 | 126
Participants | 41 | 43
Statistical Analysis 1: Comparison: DSXS 1535 vs Placebo; Test type: Superiority; p = 0.4557, Cochran-Mantel-Haenszel

2. Primary Outcome: Clinical Success in Patients With Mild to Severe Scalp Psoriasis
Description: IGA score of 0 (clear) or 1 (almost clear) with at least a 2 grades reduction from baseline
Time Frame: from baseline to study day 29
Population: Patients with mild to severe scalp psoriasis (primary analysis 2)
Measure: Count of Participants; unit: Participants
Arm/Group | DSXS 1535 | Placebo
Number analyzed (Participants) | 183 | 189
Participants | 51 | 50
Statistical Analysis 1: Comparison: DSXS 1535 vs Placebo; Test type: Superiority; p = 0.8096, Cochran-Mantel-Haenszel

3. Secondary Outcome: Clinical Success in Patients With Mild Scalp Psoriasis
Description: IGA score of 0 (clear) or 1 (almost clear) with at least a 2 grades reduction from baseline
Time Frame: from baseline to study day 29
Measure: Count of Participants; unit: Participants
Arm/Group | DSXS 1535 | Placebo
Number analyzed (Participants) | 77 | 63
Participants | 10 | 7
Statistical Analysis 1: Comparison: DSXS 1535 vs Placebo; Test type: Superiority; p = 0.7652, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | DSXS 1535 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/180 | 0/189
Serious Adverse Events (participants affected / at risk) | 0/180 | 0/189
Other Adverse Events (participants affected / at risk) | 46/180 | 43/189
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DSXS 1535 (N=180) | Placebo (N=189)
Ear discomfort (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Eye irritation (Eye disorders) | 2 (2) | 5 (5)
Eye pain (Eye disorders) | 0 (0) | 2 (2)
Eye pruritus (Eye disorders) | 2 (2) | 2 (2)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0)
Ocular discomfort (Eye disorders) | 4 (4) | 1 (1)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Application site discomfort (General disorders) | 0 (0) | 1 (1)
Application site dryness (General disorders) | 2 (2) | 1 (1)
Application site dryness (General disorders) | 1 (1) | 0 (0)
Application site pain (General disorders) | 3 (3) | 2 (2)
Application site pruritus (General disorders) | 3 (3) | 4 (4)
Asthenia (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Xerosis (General disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 2 (2)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 5 (5)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Burns third degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 7 (7) | 12 (14)
Dysmenorrhoea (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes